CLINICAL TRIAL: NCT01105637
Title: A Trial of an Augmented Exercise Program in the Prevention of Deconditioning Among Survivors of Severe Burns
Acronym: AEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HBV02-11-15-05
Record Dates: First submitted 2010-04-12; First posted 2010-04-16 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Deconditioning Among Survivors of Severe Burns
Keywords: burn injuries; exercise
MeSH Terms: conditions — Burns; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Exercise (Other)
  Interventions: Behavioral: Augmented Exercise Program

INTERVENTIONS:
Behavioral: Augmented Exercise Program — 12 week (3 x per week) exercise prescription

SUMMARY:
Burn injuries can affect how well you are able to perform daily activities. The reason this study is being done is to find out if aerobic exercise helps burn patients recover function, strength and stamina.

Participants will come to Johns Hopkins Bayview Medical Center, Burn Rehabilitation Gym for treadmill exercise sessions 3 days per week for 12 weeks. Participants will be tested for strength and stamina before the start of the 12 week program, at the end of the 12 week program, as well as 6 months, 1 year and 2 years after the end of the 12 week program.

Patients who recently suffered a burn injury and who were discharged from the hospital in the past six months may be eligible to participate.

ELIGIBILITY:
Inclusion Criteria:

* Patients who recently suffered a burn injury and who were discharged from the hospital in the past six months may be eligible to participate

Exclusion Criteria:

* History of heart-related health problems
* Foot burns

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Maximal Oxygen Consumption (VO2 max) | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J de Lateur, MD, Principal Investigator — Johns Hopkins Univeristy School of Medicine
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] de Lateur BJ, Magyar-Russell G, Bresnick MG, Bernier FA, Ober MS, Krabak BJ, Ware L, Hayes MP, Fauerbach JA. Augmented exercise in the treatment of deconditioning from major burn injury. Arch Phys Med Rehabil. 2007 Dec;88(12 Suppl 2):S18-23. doi: 10.1016/j.apmr.2007.09.003. PMID 18036976